CLINICAL TRIAL: NCT00349700
Title: An Open Prospective Controlled Trial: Efficiency of Wound Dressings Adapted to Wound Exudate and Bacterial Load in Therapy Resistant Large Sized Leg Ulcers
Brief Title: Wound Dressings Adapted to Wound Exudate and Bacterial Load in Therapy Resistant Large Sized Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-Stucker
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2006-07

CONDITIONS: Varicose Ulcer
Keywords: healing; skin; infection; wound therapy
MeSH Terms: conditions — Varicose Ulcer; Infections | interventions — Debridement; allevyn

INTERVENTIONS:
Procedure: Compression: 2 weeks four layer bandages, then stockings
Procedure: debridement
Procedure: Actisorb plus (r) + Trionic(r)/ Allevyn (r)

SUMMARY:
The purpose of the study was to investigated if modern wound dressings adapting to wound exudation and the amount of bacterial colonization can heal large therapy resistant leg ulcers which had a pre-treatment with compresses, ointments and gauze

DETAILED DESCRIPTION:
Background: Moist wound therapy of venous leg ulcers is well established by both in vitro or animal studies and studies at ulcers smaller than 20 cm². Mostly larger venous leg ulcers have a stronger exudation than smaller leg ulcers. Therefore larger ulcers exhibit apparently moist conditions also beneath simple gauze, ointments and compresses.

The purpose of the study was to investigated if modern wound dressings adapting to wound exudation and the amount of bacterial colonization can heal large therapy resistant leg ulcers which had a pre-treatment with compresses, ointments and gauze.

Patients and Methods: In an open, non-randomized prospective trial 139 consecutive patients (86 female, 53 male) with long standing (159 ± 335 weeks) large sized (> 20 cm², 53.8 ± 90.6 cm²) venous ulcers were included. The pre-treatment with compresses, ointments and gauze and two layer short stretch bandages during the time before consulting our wound outpatient department was compared to the following therapy protocol: After two weeks with four layer bandages compression stockings were applied. After a surgical debridement wound dressings were applied according to exudation (strong: calcium alginate, mean: polyurethane foam, low: hydrocolloid). Critical bacterial colonization was treated by activated charcoal cloth with sil-ver. Criteria for evaluating efficacy were healing time and reduction of ulcer size at the end of observation time.

ELIGIBILITY:
Inclusion Criteria:

* therapy resistant wounds for at least 3 months
* venous disease
* uncle pressure > 80mmHg
* wound area > 20qcm

Exclusion Criteria:

* uncle pressure <80mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139
Dates: Start 2003-01; Study Completion 2005-05

PRIMARY OUTCOMES:
the area of leg ulcers was calculated by multiplication of maximal length and width during the first visit an d at least 6 months after first visit

CONTACTS AND LOCATIONS:
Overall Officials: Peter Altmeyer, Prof. Dr., Principal Investigator — Ruhr University Bochum, Dep. Dermatology and Allergology
Locations (1):
- St. Josef Hospital, Dep. Dermatology and Allergology, Ruhr University Bochum, Bochum, Germany